CLINICAL TRIAL: NCT00019175
Title: PHASE I TRIAL IN PATIENTS WITH METASTATIC MELANOMA OF IMMUNIZATION WITH A RECOMBINANT FOWLPOX VIRUS ENCODING THE GP100 MELANOMA ANTIGEN
Brief Title: Vaccine Therapy With or Without Interleukin-2 in Treating Patients With Recurrent Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064960; NCI-96-C-0121; NCI-T94-0139N; NCT00001510 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-05-26 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2003-04

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Biological: fowlpox virus vaccine vector
Biological: gp100 antigen

SUMMARY:
RATIONALE: Vaccines made from an antigen combined with a modified virus may make the body build an immune response to kill tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill melanoma cells. Combining vaccine therapy with interleukin-2 may kill more tumor cells.

PURPOSE: Phase I trial to compare the effectiveness of vaccine therapy with or without interleukin-2 in treating patients who have recurrent metastatic melanoma that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the toxicity, immunologic reactivity, and possible therapeutic efficacy of immunization with recombinant fowlpox virus encoding the gp100 melanoma antigen administered alone or with interleukin-2 in patients with metastatic melanoma.

OUTLINE: This is a dose-escalation study. Patients receive recombinant fowlpox virus encoding the gp100 melanoma antigen (FPV-gp100) IV or intramuscularly to rotating sites or fowlpox virus encoding modified gp100 melanoma antigen IV every 2 weeks for 4 vaccinations. Treatment continues for a maximum of 2 courses in the absence of disease progression. Cohorts of 3-9 patients receive escalating doses of FPV-gp100 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients develop dose-limiting toxicity. Patients in 3 of 5 cohorts also receive interleukin-2 (IL-2) within 12 hours of FPV-gp100. One cohort receives IL-2 subcutaneously daily on days 1-5 and days 8-12. A second cohort receives low-dose IL-2 IV over 15 minutes every 8 hours on days 2-8. A third cohort receives high-dose IL-2 IV over 15 minutes every 8 hours on days 2-6. Patients in cohorts 4 and 5 receive FPV-gp100 alone and, if no response is observed after 2 courses, may receive 2 courses of IL-2 alone every 8 hours for 5 days, approximately 2 weeks apart. A separate cohort of 3-9 patients receives modified FPV-gp100. If no response is observed after 2 courses, IL-2 may be administered as in cohorts 4 and 5. Patients are followed at 28 days after the second immunization with FPV-gp100.

PROJECTED ACCRUAL: A maximum of 91 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic melanoma that has failed standard therapy Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: More than 3 months Hematopoietic: WBC greater than 3,000/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 8.0 g/dL No coagulation disorder Hepatic: Bilirubin no greater than 2.0 mg/dL AST and ALT less than 4 times normal Hepatitis B negative Renal: Creatinine no greater than 1.6 mg/dL Cardiovascular: No major cardiovascular disease Pulmonary: No major respiratory disease Other: HIV negative No other major immunologic illness No eczema No hypersensitivity to eggs No active systemic infection No psoriasis Not pregnant Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: See Disease Characteristics More than 20 days since prior therapy No concurrent steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-08

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Surgery Branch, Bethesda, Maryland, United States